CLINICAL TRIAL: NCT02645539
Title: A Clinical Study to Evaluate Ambulatory Counterpulsation for the Treatment of Advanced Heart Failure: A Feasibility Study
Brief Title: Feasibility Study of the Intravascular Ventricular Assist System (iVAS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NuPulseCV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-10001
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: Heart failure; Bridge-to-transplant; circulatory support; VAD; IABP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): All patients are treated with the intravascular ventricular assist system (iVAS).
  Interventions: Device: intravascular ventricular assist system (iVAS)

INTERVENTIONS:
Device: intravascular ventricular assist system (iVAS) — A mechanical circulatory support device using the principles of counterpulsation.
  Other Names: iVAS; Blood Pump; NuPulse

SUMMARY:
The purpose of this feasibility study is to assess the preliminary safety and clinical performance of the intravascular ventricular assist system (iVAS).

DETAILED DESCRIPTION:
This is a single-arm, non-randomized study designed to assess the preliminary safety and clinical performance of the NuPulseCV iVAS.

Data obtained from the study will be used to make device modifications, refine the patient population, and inform the design a future clinical trial suitable for assessing longer-term use in heart failure patients.

ELIGIBILITY:
Main Inclusion Criteria:

1. At least 18 years of age.
2. If female, are postmenopausal or surgically sterilized, or have a negative pregnancy test within seven (7) days of invasive testing.
3. Advanced heart failure (NYHA Class III or IV)

Main Exclusion Criteria:

1. Hypotension treated with the following medications: epinephrine, norepinephrine, vasopressin, methylene blue, phenylephrine, or angiotensin II.
2. Receiving more than two inotropes.
3. Subclavian stenosis or stent.
4. Currently receiving circulatory support including ECMO, Impella, TandemLife or equivalents; or any durable VAD.
5. Atrial fibrillation without ventricular pacing.
6. Concomitant, non-cardiac disease process with life expectancy < 1 year.
7. Significant abnormalities of the aorta, such as aneurysms, coarctation of the aorta, or an extremely tortuous aorta.
8. Severe end-organ dysfunction or failure.
9. Any other condition the heart team believes inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Survival to transplant or stroke-free survival | 30 days

SECONDARY OUTCOMES:
Number of patients who deteriorate requiring escalation of treatment | 30 days
Rate of occurrence of all adverse events | 30 days
Rate of occurrence of procedure-related adverse events | 30 days
Rate of occurrence of serious device-related adverse events | 30 days
Number of patients demonstrating improvement in NYHA Classification | 30 days
Number of patients demonstrating improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) - quality of life (QOL) | 30 days
Number of patients demonstrating improvement six minute walk test (6MWT) and two minute step test (2MST) | 30 days
Number of patients demonstrating improvement in Seattle Heart Failure Model Score | 30 days

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Advent Health, Orlando, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Saint Vincent Hospital, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Luke's Mid-America Heart Institute, Kansas City, Missouri
  - University of Nebraska, Omaha, Nebraska
  - New York University, New York, New York
  - Columbia University Medical Center / New York-Presbyterian Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - Abington Hospital - Jefferson Health, Abington, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Houston Methodist Research Institute, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah

REFERENCES:
- [Derived] Uriel N, Jeevanandam V, Imamura T, Onsager D, Song T, Ota T, Juricek C, Combs P, Lammy T, Patel-Raman S, Woolley JR, Sayer G, Milano C, Schroder J, Molina E, Grinstein J, Suarez E, Estep JD, Aggarwal S, Silvestry S, Raval N; iVAS Investigators. Clinical Outcomes and Quality of Life With an Ambulatory Counterpulsation Pump in Advanced Heart Failure Patients: Results of the Multicenter Feasibility Trial. Circ Heart Fail. 2020 Apr;13(4):e006666. doi: 10.1161/CIRCHEARTFAILURE.119.006666. Epub 2020 Apr 8. PMID 32264715